CLINICAL TRIAL: NCT01066286
Title: Genome Wide SNP Array-based Approach to Detect Micro-cytogenetic Lesions and KIT Mutation to Improve Treatment Outcomes in Patients With Core-binding Factor Positive Acute Myeloid Leukemia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Dong Hwan (Dennis) Kim/Assistant professor, Samsung Medical Center
Other Study IDs: 2009-10-069
Record Dates: First submitted 2010-02-08; First posted 2010-02-10 (Estimated); Last update posted 2010-02-10 (Estimated); Status verified 2010-02

CONDITIONS: Myeloid Leukemia
Keywords: genome wide SNP-array; micro-cytogenetic lesion; KIT mutation; core binding factor; acute myeloid leukemia; The Approval status was changed from Pending to Approved.
MeSH Terms: conditions — Leukemia, Myeloid; Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Stored bone marrow specimens of patient with core binding factor positive acute myeloid leukemia treated with chemotherapy between 1995 and 2008 at Samsung Medical Center and Hwasun Chonnam National University Hospital
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- core binding factor positive: core binding factor positive acute myeloid leukemia

SUMMARY:
Core binding factor (CBF) positive acute myeloid leukemia (AML) consist of 15% of patients in overall AML, expected to harbor a favorable prognosis. However, around a half of cases relapses. Accordingly, more sophisticated classification in CBF positive AMLs is essential to achieve further improvement in the treatment outcome. The current study is designed to evaluate CBF positive AML patients with genome-wide SNP array and KIT mutation study in CBF positive AML patients diagnosed at the Samsung Medical Center and Hwasun Chonnam National University Hospital, Korea between 1994 and 2008.

1. Construction of the CBF positive AML patient cohort: clinical database establishment (including treatment outcomes and prognosis) and extraction/storage of tumor cell DNAs from marrow samples, then processing of Affymetrix SNP array 6.0.
2. Construction of prognostic predictive model using pharmacogenomics with the results of genotypes and copy number variations (CNVs).
3. Detection of hidden microscopic cytogenetic lesions with SNP array technique, and correlation with clinical outcomes in CBF positive AML.
4. Detection of KIT, FLT3/ITD, and NPM1 gene mutation and its correlation with clinical outcomes in CBF positive AML.

The current study attempts to analyze genetic data of core binding factor (CBF) positive acute myeloid leukemia (AML) using genome wide SNP array technique with tumor DNAs collected at the time of diagnosis.

1. To detect microcytogenetic lesions and will analyze its prognostic significance
2. To analyze genome-wide genotypes and copy number variations (CNVs) using pharmacogenetic approach and will construct a prognostic predictive model
3. To detect KIT, FLT3/ITD and NPM1 mutation and evaluate its prognostic significance. The present study will establish individualized therapy for CBF positive AML, will provide a basis for molecular marker guided clinical trial in CBF positive AML.

ELIGIBILITY:
Inclusion Criteria:

* patients with core binding factor positive acute myeloid leukemia
* 18 years or older
* patients were treated with standard chemotherapy
* patients with available medical record and stored bone marrow specimen at time of diagnosis

Exclusion Criteria:

* no definive criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: core binding factor positive acute myeloid leukemia
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2010-02

PRIMARY OUTCOMES:
response rate | within 1 month after enrollment

SECONDARY OUTCOMES:
overall survival and progression-free survival | within 1 month after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Dong Hwan Kim, M.D.,Ph.D., Principal Investigator — Division of Hematology and Oncology/Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea